CLINICAL TRIAL: NCT03865290
Title: Effects of Ondansetron on Gastrointestinal Sensorimotor Dysfunctions in Diabetes Mellitus and Dyspepsia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Adil Bharucha, MBBS, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-005041; P01DK068055 (NIH)
Record Dates: First submitted 2019-02-14; First posted 2019-03-06 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Indigestion; Diabetes Mellitus
MeSH Terms: conditions — Dyspepsia; Diabetes Mellitus | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Healthy Control Ondansetron 8 mg (Experimental): Oral Ondansetron 8 mg administered in a single does dose during gastric emptying and duodenal infusion.
  Interventions: Drug: Ondansetron 8mg
- Diabetic (DM) gastroenteropathy Ondansetron 8 mg (Experimental): Oral Ondansetron 8 mg administered in a single does dose during gastric emptying and duodenal infusion.
  Oral Ondansetron 8 mg administered three times a day for weeks 3-6
  Interventions: Drug: Ondansetron 8mg
- Non-ulcer dyspepsia (NUD) Ondansetron 8 mg (Experimental): Oral Ondansetron 8 mg administered in a single does dose during gastric emptying and duodenal infusion.
  Oral Ondansetron 8 mg administered three times a day for weeks 3-6
  Interventions: Drug: Ondansetron 8mg
- Healthy Control Placebo (Placebo Comparator): Oral matched placebo administered in a single does dose during gastric emptying and duodenal infusion.
  Interventions: Drug: Placebo
- Diabetic (DM) gastroenteropathy Placebo (Placebo Comparator): Oral matched placebo administered in a single does dose during gastric emptying and duodenal infusion.
  Oral matched placebo administered three times a day for weeks 3-6
  Interventions: Drug: Placebo
- Non-ulcer dyspepsia (NUD) Placebo (Placebo Comparator): Oral matched placebo administered in a single does dose during gastric emptying and duodenal infusion.
  Oral matched placebo administered three times a day for weeks 3-6
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ondansetron 8mg — Oral Ondansetron 8 mg
  Other Names: Zofran
  Arms: Diabetic (DM) gastroenteropathy Ondansetron 8 mg; Healthy Control Ondansetron 8 mg; Non-ulcer dyspepsia (NUD) Ondansetron 8 mg
Drug: Placebo — Oral matched placebo
  Arms: Diabetic (DM) gastroenteropathy Placebo; Healthy Control Placebo; Non-ulcer dyspepsia (NUD) Placebo

SUMMARY:
Researchers are trying to understand why people with indigestion and diabetes mellitus have gastrointestinal symptoms and in particular to understand whether symptoms are related to increased sensitivity to nutrients in the small intestine. As part of this investigation, a medication called ondansetron will also be studied to determine its effects on gastrointestinal function and associated symptoms.

DETAILED DESCRIPTION:
The primary objectives of this study are to evaluate the effects of ondansetron, on symptoms (i) during a gastric emptying study, (ii) during enteral lipid infusion and (iii) in daily life.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant, non-breastfeeding female volunteers;
* 18-75 years old;
* Able to provide written informed consent before participating in the study
* Able to communicate adequately with the investigator and to comply with the requirements for the entire study; including the willingness and ability to consume the components of the test meals
* Symptoms of dyspepsia (i.e., early satiety, postprandial discomfort, nausea, vomiting, regurgitation)
* Patients in the DM group will also require Type 1 or 2 DM of ≥ 3 years duration; in patients with type 2 DM, the dyspepsia symptoms should have begun or worsened after DM was diagnosed

Exclusion Criteria:

* Major abdominal surgery (i.e., appendectomy, cholecystectomy, tubal ligation, hysterectomy, herniorrhaphy, and limited colonic resection are permissible)
* Clinical evidence (including physical exam and EKG) of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric or other disease that may interfere with the objectives of the study and/or pose safety concerns
* Current use of opiates, alpha adrenergic agonists, metoclopramide, monoamine oxidase inhibitors, more than one serotonergic medication, and high doses of anticholinergic agents (eg, amitriptyline greater than 50 mg daily). If medically safe, these drugs may be discontinued for four half lives prior to study assessments.
* Treatment with GLP-1 agonists and amlyin which cause vagal blockade and may affect central processing of pain
* Bleeding or clotting disorders or medications that increase risk of bleeding from mucosal biopsies
* Positive tissue transglutaminase antibodies (TTG),
* Pregnant or breast-feeding females
* Known intolerance or allergy to eggs
* Poor peripheral venous access, if central venous access is not available
* Any other condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study
* History of Long QT Syndrome or prolonged QT interval (i.e., corrected QT interval > 480 ms)
* Current symptoms of a functional gastrointestinal disorder assessed by questionnaire
* Severe vomiting that would preclude tube placement or participation in the study
* Structural cause for symptoms by endoscopy within the past 12 months
* Patients with gastric pacemakers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in severity of symptoms during enteral infusion | baseline, every 15 minutes up to 8 hours
  Visual analog scale (VAS) used to measure the change in symptom severity with a scale of 0=absent, 1=light, 2=moderate, 3=severe, 4=intolerable
Change in severity of symptoms during gastric emptying study | baseline, every 15 minutes up to 2 hours
  Visual analog scale (VAS) used to measure the change in symptom severity with a scale of 0=absent, 1=light, 2=moderate, 3=severe, 4=intolerable
Change in severity of daily symptoms | Baseline, daily for six weeks
  Gastroparesis Cardinal Symptom Index - Daily Diary (GCSI-DD) used to measure the change in symptoms severity with a scale of 0=none, 1= very mild, 2=mild,3=moderate, 4=severe, 5= very severe
Change in severity of gastrointestinal symptoms | Baseline, 2 weeks, 6 weeks
  Gastrointestinal Disorders - Symptom Severity Index (PAGI-SYM) used to measure the change in symptoms severity with a scale of 0=none, 1= very mild, 2=mild,3=moderate, 4=severe, 5= very severe
Change in severity of gastrointestinal symptoms effect on Quality of Life | Baseline, 2 weeks, 6 weeks
  Gastrointestinal Disorders - Quality of Life and Well-Being (PAGI-QOL) used to measure the change in symptoms severity with a scale of 0=none, 1= very mild, 2=mild,3=moderate, 4=severe, 5= very severe
Change in effect of Gastrointestinal symptoms on Quality of Life | Baseline
  Nepean Dyspepsia Index used to measure symptoms severity with a scale of 0=none, 1= very mild, 2=mild,3=moderate, 4=severe, 5= very severe

SECONDARY OUTCOMES:
Glucose level | baseline, approximately 60-120 minutes
  Compare the changes in glucose level during a lipid infusion
Insulin level | baseline, approximately 60-120 minutes
  Compare the changes in insulin level during a lipid infusion
C-peptide level | baseline, approximately 60-120 minutes
  Compare the changes in C-peptide level during a lipid infusion
Glucagon-like Peptide 1 (GLP-1) | baseline, approximately 60-120 minutes
  Compare the changes in Glucagon-like Peptide 1 (GLP-1) level during a lipid infusion
Cholecystokinin (CCK) | baseline, approximately 60-120 minutes
  Compare the changes in Cholecystokinin (CCK) level during a lipid infusion
Ghrelin | baseline, approximately 60-120 minutes
  Compare the changes in Ghrelin level during a lipid infusion
Peptide YY (PYY) | baseline, approximately 60-120 minutes
  Compare the change in Peptide YY (PYY) level during a lipid infusion
Plasma | baseline, approximately 60-120 minutes
  Compare the change in plasma level during a lipid infusion
Effect of gastrointestinal symptoms on Quality of Life - Nepean Dyspepsia index | Baseline
  Score is derived from 25 items pertaining to QOL
Severity of gastrointestinal symptoms - Nepean Dyspepsia index | Baseline
  Nepean Dyspepsia Index is used to measure symptom severity with a scale of 0=none, 1= very mild, 2=mild,3=moderate, 4=severe, 5= very severe

CONTACTS AND LOCATIONS:
Overall Officials: Adil E Bharucha, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No